CLINICAL TRIAL: NCT05711810
Title: Cardiac Transfer of SARS-CoV-2 Spike Protein Circulation Techniques - Medicine Induced Hemodialysis on "Vaccinated" Immune Attacks
Brief Title: Medicine-induced Cardiac Hemodialysis on COVID-19
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yang I. Pachankis (Individual)
Responsible Party: Sponsor-Investigator, Yang I. Pachankis, Principal Investigator, Pachankis, Yang I., M.D.
Organization: Pachankis, Yang I., M.D. (Individual)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SARSCoVVaxPoison
Record Dates: First submitted 2023-01-12; First posted 2023-02-03 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Severe Acute Respiratory Syndrome-related Coronavirus; Renal Dialysis; Vaccines; Myocarditis Allergic; Infection Viral
Keywords: immune infection; neural infection; spike 2 protein; poison; SARS-CoV-2; precarditis
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; Virus Diseases | interventions — Nifedipine; low mobility group protein 160, rat; Enalapril; Lansoprazole; Metoprolol; coenzyme Q10; alpha-Tocopherol; Docosahexaenoic Acids; Duloxetine Hydrochloride; Capsules; Superoxide Dismutase

STUDY DESIGN:
Intervention Model Description: The crossover model intervenes on the precarditis and myocarditis happenings on the patient, and evaluates the cause of the symptoms. Basic medicines are tested against the pathogens with the immune responses of the patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Experiment Participant (Experimental): COVID-19 recombined vaccinated, 3 dose, no intervention. Nifedipine, oral, 30 mg per day for 2 days, active comparative. Angiotensin-converting enzyme inhibitor, oral, gradually increase to 20 mg per day at night.
  Beta blocker, oral, 23.75 - 95 mg per day in the morning. Proton-pump inhibitor, oral, 30 mg per day. Duloxetine hydrochloride, oral, placebo, 20 mg per day before sleep. Acetaminophen (sham comparator), oral, 250 mg four times per day for 8 days. Cefuroxime (sham comparator), oral, 100 mg twice per day for 6 days. Papaverine, oral, low-dosage in coughing pills for 4 days. Superoxide Dismutase (active comparator), oral, to be introduced. Bafilomycin A1 (active comparator), oral, 100 ug per kilogram per day, unlikely to be introduced for lack of funding.
  Interventions: Drug: Nifedipine 30 MG; Diagnostic Test: Kangzhu BPCB0A-3A; Behavioral: Low Mobility; Drug: Enalapril Maleate 10Mg Tab; Drug: Lansoprazole 30Mg Ec Cap; Drug: Metoprolol Succinate; Dietary Supplement: Coenzyme Q10; Dietary Supplement: d-alpha tocopherol acetate; Dietary Supplement: Omega-3; Drug: Duloxetine Hydrochloride 20 MG Oral Capsule, Delayed Release; Drug: Superoxide Dismutase

INTERVENTIONS:
Drug: Nifedipine 30 MG — Due to initial availability of drugs and the intensities of the patient's symptoms, Nifedipine was used for initial intervention in preventing acute myocarditis from happening.
  Other Names: Nifedipine Control-release Tablets
Diagnostic Test: Kangzhu BPCB0A-3A — The diagnostic test has been used to confirm objective parameters to guide the intervention drug dosages and accessing the risks in sudden death and long term adverse effects.
  Other Names: Heart Monitor
Behavioral: Low Mobility — The behavioral intervention aimed at reducing the risks of sudden and strong blood flows in the patient's system.
Drug: Enalapril Maleate 10Mg Tab — The intervention aims to reduce the vein flows in Diastolic Blood Pressure, and the risks in blood clot formation and internal vein scratch bleeding.
Drug: Lansoprazole 30Mg Ec Cap — The intervention aims to server the allergy-inducing proteins to induce renal hemodialysis.
Drug: Metoprolol Succinate — Metoprolol Succinate is used to control the cardiac artery flow amounts and stabilize the patient's heart rate.
Dietary Supplement: Coenzyme Q10 — 200 mg per day is used for supplement with the cardiac interventions.
Dietary Supplement: d-alpha tocopherol acetate — The 268 mg twice per day dietary healthcare is the patient's usual daily use.
Dietary Supplement: Omega-3 — The 900 mg twice per day dietary healthcare is the patient's usual daily use.
Drug: Duloxetine Hydrochloride 20 MG Oral Capsule, Delayed Release — Duloxetine hydrochloride is used for the patient's neurodiverse conditions.
  Other Names: Neurodiverse
Drug: Superoxide Dismutase — Superoxide Dismutase is used to substitute the missing of antiviral drugs.

SUMMARY:
The clinical trial studies the human pathogen of SARS-CoV-2, with a specificity in the circulating Spike 2 protein in the human system. The clinical trial hypothesizes that SARS-CoV-2 human pathogen arises from immune attacks, underlying the severe physiological symptoms that can be lethal. It further hypothesizes that the vaccines do not deal with the Spike 2 protein that causes the immune attacks.

ELIGIBILITY:
Inclusion Criteria:

* No mRNA vaccinated poisoning have been included currently, but scientific evidence suggest the methods of vaccination are irrelevant to the conditions. It is theorized that the more advanced the vaccine production technology, the deeper the poisoning.

Exclusion Criteria:

* healthy individuals with no myocarditis or unvaccinated without infection by SARS-CoV series
* persons with diabetes (Paxlovid and PrEP treatments can be applied according to availability)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-12 (Actual)

PRIMARY OUTCOMES:
Heart Rate | 1 day
  The heart rate is monitored daily, and the primary goal is to stabilize the patient's heart rate.
Electrocardiogram | 20 days
  Electrocardiogram reflects the blood pressure management on the patient's health outcome and potential risks.
Platelet Distribution | 10 days
  Platelet distribution is measured to determine the viral induced blood-borne pathogen in the physiological responses of the patient.
Mean Platelet Volume | 10 days
  MPV is measured to determine the risks in blood clot and internal vein scratches in the patient.
Eosinophil Absolute Number | 10 days
  Eosinophil Absolute Number is measured to determine the intensities of infection in the patient.
Basophil Absolute Number | 10 days
  Basophil Absolute Number is measured on the counteraction of the patient's immune system integrities against the rapid acidification of the viral infection.

SECONDARY OUTCOMES:
Cardiac Enzymes | 10 days
  Cardiac enzymes are measured to locate and eliminate the symptoms' causes, identify potential health risks, and to determine if subsidiary treatments are needed.

CONTACTS AND LOCATIONS:
Locations (1):
- Residential Address, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The emergent intervention started with the PI's research into the virology and post-vaccination adverse effects. The plan was improvised and adjusted accordingly. Statistical analysis was mainly physiological with relation to the virological inductions from the patient's symptomatic responses.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The first 20 days of data have been uploaded on Zenodo, and significant results and monitoring data will be updated accordingly.
Access Criteria: The data is openly available on Zenodo. The hospital facility and personnel involved for prescription drugs and tests are deidentified.
URL: https://doi.org/10.5281/zenodo.7588613

REFERENCES:
- [Background] Liu X, Mostafavi H, Ng WH, Freitas JR, King NJC, Zaid A, Taylor A, Mahalingam S. The Delta SARS-CoV-2 Variant of Concern Induces Distinct Pathogenic Patterns of Respiratory Disease in K18-hACE2 Transgenic Mice Compared to the Ancestral Strain from Wuhan. mBio. 2022 Jun 28;13(3):e0068322. doi: 10.1128/mbio.00683-22. Epub 2022 Apr 14. PMID 35420469
- [Background] Wu Zhang X, Leng Yap Y. Structural similarity between HIV-1 gp41 and SARS-CoV S2 proteins suggests an analogous membrane fusion mechanism. Theochem. 2004 May;677(1):73-76. doi: 10.1016/j.theochem.2004.02.018. Epub 2004 Apr 2. PMID 32287546
- [Background] Hu B, Guo H, Zhou P, Shi ZL. Characteristics of SARS-CoV-2 and COVID-19. Nat Rev Microbiol. 2021 Mar;19(3):141-154. doi: 10.1038/s41579-020-00459-7. Epub 2020 Oct 6. PMID 33024307
- [Background] Xavier LL, Neves PFR, Paz LV, Neves LT, Bagatini PB, Timmers LFSM, Rasia-Filho AA, Mestriner RG, Wieck A. Does Angiotensin II Peak in Response to SARS-CoV-2? Front Immunol. 2021 Jan 14;11:577875. doi: 10.3389/fimmu.2020.577875. eCollection 2020. PMID 33519802
- [Background] Ortiz-Guerrero G, Amador-Munoz D, Calderon-Ospina CA, Lopez-Fuentes D, Nava Mesa MO. Proton Pump Inhibitors and Dementia: Physiopathological Mechanisms and Clinical Consequences. Neural Plast. 2018 Mar 21;2018:5257285. doi: 10.1155/2018/5257285. eCollection 2018. PMID 29755512
- [Background] Tabares L, Betz B. Multiple functions of the vesicular proton pump in nerve terminals. Neuron. 2010 Dec 22;68(6):1020-2. doi: 10.1016/j.neuron.2010.12.012. PMID 21172605
- [Background] Goldstein FC, Steenland K, Zhao L, Wharton W, Levey AI, Hajjar I. Proton Pump Inhibitors and Risk of Mild Cognitive Impairment and Dementia. J Am Geriatr Soc. 2017 Sep;65(9):1969-1974. doi: 10.1111/jgs.14956. Epub 2017 Jun 7. PMID 28590010
- [Background] Poea-Guyon S, Ammar MR, Erard M, Amar M, Moreau AW, Fossier P, Gleize V, Vitale N, Morel N. The V-ATPase membrane domain is a sensor of granular pH that controls the exocytotic machinery. J Cell Biol. 2013 Oct 28;203(2):283-98. doi: 10.1083/jcb.201303104. PMID 24165939
- [Background] Wang D, Hiesinger PR. The vesicular ATPase: a missing link between acidification and exocytosis. J Cell Biol. 2013 Oct 28;203(2):171-3. doi: 10.1083/jcb.201309130. PMID 24165933
- [Background] Glebov OO. Understanding SARS-CoV-2 endocytosis for COVID-19 drug repurposing. FEBS J. 2020 Sep;287(17):3664-3671. doi: 10.1111/febs.15369. Epub 2020 Jun 2. PMID 32428379
- [Background] Ragia G, Manolopoulos VG. Inhibition of SARS-CoV-2 entry through the ACE2/TMPRSS2 pathway: a promising approach for uncovering early COVID-19 drug therapies. Eur J Clin Pharmacol. 2020 Dec;76(12):1623-1630. doi: 10.1007/s00228-020-02963-4. Epub 2020 Jul 21. PMID 32696234
- [Background] Cure E, Cumhur Cure M. Angiotensin-converting enzyme inhibitors and angiotensin receptor blockers may be harmful in patients with diabetes during COVID-19 pandemic. Diabetes Metab Syndr. 2020 Jul-Aug;14(4):349-350. doi: 10.1016/j.dsx.2020.04.019. Epub 2020 Apr 15. PMID 32311651
- [Background] Duwal S, Schutte C, von Kleist M. Pharmacokinetics and pharmacodynamics of the reverse transcriptase inhibitor tenofovir and prophylactic efficacy against HIV-1 infection. PLoS One. 2012;7(7):e40382. doi: 10.1371/journal.pone.0040382. Epub 2012 Jul 11. PMID 22808148
- [Background] Bradley BT, Bryan A, Fink SL, Goecker EA, Roychoudhury P, Huang ML, Zhu H, Chaudhary A, Madarampalli B, Lu JYC, Strand K, Whimbey E, Bryson-Cahn C, Schippers A, Mani NS, Pepper G, Jerome KR, Morishima C, Coombs RW, Wener M, Cohen S, Greninger AL. Anti-SARS-CoV-2 Antibody Levels Measured by the AdviseDx SARS-CoV-2 Assay Are Concordant with Previously Available Serologic Assays but Are Not Fully Predictive of Sterilizing Immunity. J Clin Microbiol. 2021 Aug 18;59(9):e0098921. doi: 10.1128/JCM.00989-21. Epub 2021 Aug 18. PMID 34165323
- [Background] Graham RL, Baric RS. Recombination, reservoirs, and the modular spike: mechanisms of coronavirus cross-species transmission. J Virol. 2010 Apr;84(7):3134-46. doi: 10.1128/JVI.01394-09. Epub 2009 Nov 11. PMID 19906932
- [Background] Pham AQ, Xu LH, Moe OW. Drug-Induced Metabolic Acidosis. F1000Res. 2015 Dec 16;4:F1000 Faculty Rev-1460. doi: 10.12688/f1000research.7006.1. eCollection 2015. PMID 26918138
- [Background] Fischer W, Giorgi EE, Chakraborty S, Nguyen K, Bhattacharya T, Theiler J, Goloboff PA, Yoon H, Abfalterer W, Foley BT, Tegally H, San JE, de Oliveira T; Network for Genomic Surveillance in South Africa (NGS-SA); Gnanakaran S, Korber B. HIV-1 and SARS-CoV-2: Patterns in the evolution of two pandemic pathogens. Cell Host Microbe. 2021 Jul 14;29(7):1093-1110. doi: 10.1016/j.chom.2021.05.012. Epub 2021 Jun 3. PMID 34242582
- [Background] Dilip KG. Poison as Discussed by Susruta, The Father of Surgery. Biomedical Science and Clinical Research. 2022; 1(1): 18-20.
- [Background] Yonker LM, Swank Z, Bartsch YC, Burns MD, Kane A, Boribong BP, Davis JP, Loiselle M, Novak T, Senussi Y, Cheng CA, Burgess E, Edlow AG, Chou J, Dionne A, Balaguru D, Lahoud-Rahme M, Arditi M, Julg B, Randolph AG, Alter G, Fasano A, Walt DR. Circulating Spike Protein Detected in Post-COVID-19 mRNA Vaccine Myocarditis. Circulation. 2023 Mar 14;147(11):867-876. doi: 10.1161/CIRCULATIONAHA.122.061025. Epub 2023 Jan 4. PMID 36597886
- [Background] Yang IP. Public health equity in information asymmetry - phenomenological studies upon SARS-CoV-2 super- virus mutation. International Physical Medicine & Rehabilitation Journal. 2023; 8(1): 14-18.
- See also: B6.Cg-Tg(K18-ACE2)2Prlmn/J — http://www.jax.org/strain/034860
- See also: Proton Pump Inhibitors — http://patient.info/digestive-health/indigestion-medication/proton-pump-inhibitors
- See also: SARS CoV 2 Spike Antibody, IgG — http://testguide.labmed.uw.edu/view/NCVIGQ?tabs=no
- See also: Angiotensin Converting Enzyme Inhibitors (ACEI) — http://www.ncbi.nlm.nih.gov/books/NBK431051/
- See also: Low basophil count in the blood — http://www.mrlabtest.com/low-basophils-blood.htm
- See also: Normal basophil count in the blood — http://www.mrlabtest.com/normal-basophils-blood.htm
- Available data/document: Clinical Study Report: 10.5281/zenodo.7534361 — https://doi.org/10.5281/zenodo.7534361 — The local hospital and medicare information are deidentified for their protection.